CLINICAL TRIAL: NCT06972225
Title: Follow-up of MACE in Patients Treated With Drug-eluting Balloons Between 2010 and 2025; a Retrospective Study With Prospective Follow-up From an Institutional Database: EASY-drug-eluting Balloons
Brief Title: Restrospective Analysis of MACE in Patients Treated With Drug-elluting Balloons.
Acronym: EASY-DEB
Status: Not yet recruiting | Type: Observational
Sponsor: Olivier F. Bertrand (Other)
Responsible Party: Sponsor-Investigator, Olivier F. Bertrand, MD, PhD, Laval University
Organization: Laval University (Other)
Other Study IDs: EASY-DEB
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Coronary Arterial Disease (CAD); Restenosis, Coronary; Bifurcation Coronary Disease
MeSH Terms: conditions — Coronary Restenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DEB
  Interventions: Device: DEB

INTERVENTIONS:
Device: DEB — Use of DEB to treat coronary lesions

SUMMARY:
Retrospective analysis of data collected in an institutional database of coronary interventions with use of drug-eluting balloons, with a prospective follow-up for major adverse cardiovascular events and living status.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>=18 years of age)
* Who underwent a coronary angioplasty with drug-eluting balloon between January 2010 and December 2025
* Identified in the institutional procedure database

Exclusion Criteria:

* Incomplete or non-available data on the post-procedural clinical follow-up
* Procedures where other devices were used in combination with drug-eluting balloons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients registered in the institutional procedural database who underwent a coronary angioplasty with drug-eluting balloons exclusively between January 2010 and December 2025.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2035-12 (Estimated); Study Completion 2036-03 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events | within 10 years of inclusion
  defined as:
  * Cardiovascular death
  * Myocardial infarction
  * Target vessel revascularization
  * Cerebrovascular event
  * Hospitalization due to heart failure

CONTACTS AND LOCATIONS:
Locations (1):
- IUCPQ, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Scheller B, Hehrlein C, Bocksch W, Rutsch W, Haghi D, Dietz U, Bohm M, Speck U. Treatment of coronary in-stent restenosis with a paclitaxel-coated balloon catheter. N Engl J Med. 2006 Nov 16;355(20):2113-24. doi: 10.1056/NEJMoa061254. Epub 2006 Nov 13. PMID 17101615
- [Background] Giacoppo D, Saucedo J, Scheller B. Coronary Drug-Coated Balloons for De Novo and In-Stent Restenosis Indications. J Soc Cardiovasc Angiogr Interv. 2023 Mar 30;2(3):100625. doi: 10.1016/j.jscai.2023.100625. eCollection 2023 May-Jun. PMID 39130710
- [Background] Jeger RV, Eccleshall S, Wan Ahmad WA, Ge J, Poerner TC, Shin ES, Alfonso F, Latib A, Ong PJ, Rissanen TT, Saucedo J, Scheller B, Kleber FX; International DCB Consensus Group. Drug-Coated Balloons for Coronary Artery Disease: Third Report of the International DCB Consensus Group. JACC Cardiovasc Interv. 2020 Jun 22;13(12):1391-1402. doi: 10.1016/j.jcin.2020.02.043. Epub 2020 May 27. PMID 32473887